CLINICAL TRIAL: NCT00564733
Title: FDG-PET Based Chemotherapy Selection for Metastatic Non-Small Cell Lung Cancer
Brief Title: FDG-Labeled PET Scan in Planning Chemotherapy in Treating Patients With Stage IIIB or IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Keith D Eaton, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6566; NCI-2010-00606 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 5R21CA123866-02 (NIH)
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Malignant Pleural Effusion; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Pleural Effusion, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Docetaxel; Gemcitabine; Paclitaxel; Taxes; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Patients undergo FDG PET/CT (fludeoxyglucose F 18 positron emission tomography/computed tomography) scan between days 18-21. The FDG PET/CT is an imaging biomarker analysis. Patients that are responding to treatment receive paclitaxel IV and carboplatin IV on day 1. Treatment repeats every 3 weeks for up to 3 additional courses in the absence of disease progression or unacceptable toxicity.Patients that are not responding to chemotherapy per FDG PET then receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and docetaxel IV over 1 hour on day 8. Treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Non-responding patients undergo an additional FDG PET/CT scan between days 18-21 of course 2.
  Interventions: Drug: carboplatin; Drug: docetaxel; Drug: gemcitabine hydrochloride; Drug: paclitaxel; Procedure: computed tomography; Procedure: positron emission tomography; Radiation: fludeoxyglucose F 18; Other: imaging biomarker analysis

INTERVENTIONS:
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Procedure: computed tomography — Undergo FDG PET/CT
  Other Names: tomography, computed
Procedure: positron emission tomography — Undergo FDG PET/CT
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Radiation: fludeoxyglucose F 18 — Given IV
  Other Names: 18FDG; FDG
Other: imaging biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well fludeoxyglucose F 18 (FDG)-labeled positron emission tomography (PET) scan works in planning chemotherapy in treating patients with stage IIIB or IV non-small cell lung cancer (NSCLC). Drugs used in chemotherapy, such as paclitaxel, carboplatin, gemcitabine hydrochloride, and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Diagnostic imaging procedures, such as FDG-labeled PET scan, may help in guiding chemotherapy and allow doctors to plan better treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the response rate in patients who do not demonstrate an early response to carboplatin/paclitaxel as determined by FDG-PET ("initial non-responders") who are subsequently treated with three additional courses of docetaxel/gemcitabine.

SECONDARY OBJECTIVES:

I. Evaluate the ability of FDG-PET to predict response to therapy as measured by computed tomography (CT).

II. Evaluate the early and late changes in tumor FDG uptake (change in standardized uptake value [SUV]) in all patients and correlate with overall survival (OS).

OUTLINE: All patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 1. Patients undergo FDG-PET/CT scan between days 18-21.

Patients are then assigned to 1 of 2 treatment groups.

GROUP I (Responders): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 3 additional courses in the absence of disease progression or unacceptable toxicity.

GROUP II (Initial non-responders): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and docetaxel IV over 1 hour on day 8. Treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients undergo FDG-PET/CT scan between days 18-21 of course 2.

After completion of study treatment, patients are followed up at days 81-84 and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed NSCLC; patients must have stage IIIB with malignant pleural effusion or with nodal disease so extensive that it is not amenable to radiotherapy with curative intent, or stage IV disease, as defined by the American Joint Committee on Cancer (AJCC) cancer staging handbook, 6th Edition (2002)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (>= 10 mm with spiral CT scan); patients' baseline FDG-PET scan must demonstrate a target lesion with SUV >= 2 x background and SUV > 3
* All patients must not have received treatment with conventional cytotoxic chemotherapy for NSCLC; patients may have had prior radiotherapy or may have been treated with the epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKI) (i.e. erlotinib or gefitinib); one week must have elapsed after discontinuation, prior to the initial PET scan for patients previously treated with a TKI; patients who receive radiotherapy must have recovered from the side effects of therapy (except alopecia) and have measurable disease (target lesion) outside of the radiation field
* Life expectancy >= 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) =< 2 x institutional ULN (< 5 x ULN for patients with liver metastases)
* Creatinine =< 1.5 x ULN OR creatinine clearance >= 40 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have baseline FDG-PET and CT scans performed at the University of Washington (UW)/Seattle Cancer Care Alliance (SCCA) within two weeks from the start of chemotherapy
* Asymptomatic patients with clinically stable brain metastases (treated or untreated) are allowed
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) throughout treatment and for 30 days following the last dose of chemotherapy
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have received EGFR TKI (i.e. erlotinib or gefitinib) within one week prior to entering the study
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition agents used in the study
* Inability or unwillingness to take corticosteroids, which are required pre-medications for the chemotherapies in this trial
* Diabetes requiring insulin for management
* Patients must weigh less than 400 lbs
* Patients with post-obstructive pneumonia or lobar collapse
* Significant neuropathy (common toxicity criteria [CTC] grade > 2), as both the paclitaxel and docetaxel have potential for neurotoxicity
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women
* Patients with a detectable second malignancy are excluded, as this could confound tumor evaluation and affect patient survival
* Patients who are likely to need palliative radiation therapy for painful bony metastases, impending fractures, or hemoptysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-10; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Eaton, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Patients undergo FDG PET/CT scan between days 18-21. Patients that are responding to treatment receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 3 additional courses in the absence of disease progression or unacceptable toxicity.Patients then receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and docetaxel IV over 1 hour on day 8. Treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients undergo FDG PET/CT scan between days 18-21 of course 2.
  carboplatin: Given IV
  docetaxel: Given IV
  gemcitabine hydrochloride: Given IV
  paclitaxel: Given IV
  computed tomography: Undergo FDG PET/CT
  positron emission tomography: Undergo FDG PET/CT
  fludeoxyglucose F 18: Given IV
  imaging biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Chemotherapy
Started | 55
Completed | 46
Not Completed | 9
Not completed — Withdrawal by Subject | 4
Not completed — Ineligible | 5

BASELINE CHARACTERISTICS:
Population: All patients that signed consent and received at least one dose of chemotherapy.
Arm/Group | Chemotherapy
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 18
Age, Continuous [Mean (Full Range); unit: years] | 60 [48 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 22
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Patients That Achieve a CR or PR)
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: At the end of 4 cycles of treatment, up to 24 weeks.
Population: All patients that signed consent and received at least one cycle of chemotherapy.
Measure: Number; unit: participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 46
participants | 13

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing the informed consent through 30 days after the final dose of chemotherapy, up to 24 weeks.
Description: Only grade 3 and higher adverse events or adverse events that led to a dose reduction or dose delay were captured. Hospitalizations related to disease progression were not captured as serious adverse events.
Arm/Group | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 3/46
Other Adverse Events (participants affected / at risk) | 20/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=46)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Neutropenia (Investigations) | 1 (1)
acute renal insufficiency (Renal and urinary disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=46)
Increased ALT (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Fatigue (General disorders) | 6 (6)
Fever (General disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (4)
Lymphocyte count decreased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (3)
Pain- NOS (Musculoskeletal and connective tissue disorders) | 5 (5)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Thrombocytopenia (Investigations) | 7 (8)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No